CLINICAL TRIAL: NCT07172451
Title: Efficacy and Safety of Balanced Gelatin Solution for Fluid Infusion in Sepsis Patients Undergoing Emergency Abdominal Surgery: A Multicenter, Adaptive Designed, Randomized Controlled Trial
Brief Title: Gelaspan vs Crystalloid Therapy in Sepsis
Acronym: SPACES
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: B. Braun Medical International Trading Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZSANES.B2025-465R; Ethics Approval No. B2025-465R (Other: Ethics Committee of Zhongshan Hospital, Fudan University)
Record Dates: First submitted 2025-09-03; First posted 2025-09-15 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Sepsis; Intra-Abdominal Infections
Keywords: Balanced gelatin solution; Succinylated gelatin; Crystalloid; Ringer's acetate; Fluid resuscitation; Goal-directed fluid therapy; Emergency abdominal surgery; Microcirculation; Hemodynamic stabilization; SOFA score; Lactate clearance; Randomized controlled trial
MeSH Terms: conditions — Sepsis; Intraabdominal Infections | interventions — Ringer's acetate

STUDY DESIGN:
Intervention Model Description: This is a prospective, multicenter, double-blind, randomized controlled clinical trial with a parallel assignment design. Eligible patients will be randomized in a 1:1 ratio to receive either balanced gelatin solution or crystalloid solution as the primary resuscitation fluid during emergency abdominal surgery for sepsis. Randomization is stratified by baseline lactate level (≤4 vs. >4 mmol/L) using a central dynamic allocation system.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This trial uses a double-blind design. Participants, treating clinicians (care providers), investigators, and outcomes assessors are all blinded to treatment allocation. Study fluids (balanced gelatin vs. crystalloid) are packaged in identical opaque containers by an independent coordinator who is not involved in patient care or outcome assessment. Randomization and labeling are performed centrally, and only the data monitoring committee has access to unblinded allocation if required for patient safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Balanced Gelatin Solution (Experimental): Patients randomized to the balanced gelatin group will receive balanced gelatin solution (4% succinylated gelatin in a balanced crystalloid carrier) as the primary resuscitation fluid during emergency abdominal surgery for sepsis. Fluid administration follows a goal-directed protocol guided by stroke volume monitoring. The maximum total volume of balanced gelatin is limited to 30 mL/kg (ideal body weight) within the intraoperative and first 24-hour postoperative period. If the limit is reached, additional resuscitation will be performed with balanced crystalloid solution.
  Interventions: Drug: Balanced Gelatin Solution
- Crystalloid Solution (Active Comparator): Patients randomized to the crystalloid group will receive acetate Ringer's solution as the sole resuscitation fluid during emergency abdominal surgery for sepsis, according to the same goal-directed protocol guided by stroke volume monitoring. No gelatin solution will be administered in this group. The total volume of crystalloid infusion is not limited.
  Interventions: Drug: Acetate Ringer's Solution

INTERVENTIONS:
Drug: Balanced Gelatin Solution — Balanced gelatin solution (4% succinylated gelatin in a balanced crystalloid carrier). Administered as resuscitation fluid in patients with sepsis undergoing emergency abdominal surgery. Infusion follows a stroke volume-guided, goal-directed fluid therapy protocol. The total dose is limited to 30 mL/kg (ideal body weight) during the intraoperative period and the first 24 postoperative hours. If the maximum dose is reached, additional resuscitation is provided with balanced crystalloid solution.
  Other Names: Succinylated Gelatin 4%; Gelatin Infusion; Gelaspan
  Arms: Balanced Gelatin Solution
Drug: Acetate Ringer's Solution — Acetate Ringer's solution, a balanced crystalloid, administered as the sole resuscitation fluid in patients with sepsis undergoing emergency abdominal surgery. Fluid therapy follows the same stroke volume-guided, goal-directed protocol as the experimental arm. There is no upper limit for the total volume of crystalloid infusion during the intraoperative and first 24 postoperative hours.
  Other Names: Balanced Crystalloid Solution; Ringer's Acetate
  Arms: Crystalloid Solution

SUMMARY:
The goal of this randomized clinical trial is to evaluate whether balanced gelatin solution is more effective and safe than balanced crystalloid solution for perioperative fluid management in adults with sepsis undergoing emergency abdominal surgery. Sepsis often causes severe fluid loss from the bloodstream into tissues, leading to low blood pressure, impaired organ function, and the need for urgent fluid resuscitation. Balanced gelatin, a colloid solution, may help maintain intravascular volume more effectively than crystalloid alone.

In this study, participants are randomly assigned in a 1:1 ratio to receive either balanced gelatin or Ringer's acetate during surgery and in the first 24 hours afterward. All patients receive standardized anesthesia care, goal-directed fluid therapy, and protocolized use of vasoactive drugs. The main questions the study aims to answer are:

* Does balanced gelatin reduce positive fluid balance within 24 hours after surgery?
* Does it improve hemodynamic stability during the early postoperative period?
* What effects does balanced gelatin have on kidney function, microcirculation, postoperative recovery, and other clinical outcomes?

Participants will be followed throughout hospitalization and contacted again on postoperative day 28 and day 90 to assess survival, complications, and health-related quality of life. The trial is double-blind, meaning that patients, clinicians, and outcome assessors do not know which fluid is being used. An independent Data and Safety Monitoring Board will oversee patient safety during the study.

The findings of this trial are expected to provide important evidence to guide perioperative fluid resuscitation strategies for septic patients undergoing emergency surgery.

DETAILED DESCRIPTION:
Study Background Sepsis is a life-threatening syndrome caused by a dysregulated host response to severe infection, which can rapidly progress to septic shock, multiple organ dysfunction, and death.Despite advances in recognition and treatment in recent years, sepsis remains a major global health challenge, with overall mortality rates still ranging from 18% to 30%.Pathophysiologically, sepsis is characterized by increased capillary permeability and vasodilation, resulting in substantial fluid extravasation into the interstitial space, tissue edema, and intravascular volume depletion. These changes lead to inadequate tissue perfusion, impaired oxygen delivery, and ultimately organ dysfunction. Therefore, timely and appropriate fluid resuscitation remains one of the most fundamental and essential components of sepsis management. Individualized, goal-directed fluid therapy aims to improve systemic perfusion while minimizing the risks associated with fluid overload.

In 2001, Rivers et al. introduced the concept of early goal-directed therapy (EGDT), demonstrating significant mortality reduction (30.5% vs 45%) in patients with severe sepsis and septic shock.This finding prompted widespread adoption of early aggressive fluid resuscitation. However, three large multicenter trials published between 2014 and 2015 (ARISE, ProCESS, and ProMISe) later found no significant mortality differences between EGDT and usual care (approximately 18-25%).These results suggested that with improvements in routine clinical practice, contemporary usual care may already include adequate hemodynamic optimization.

Based on this evidence, the 2016 Surviving Sepsis Campaign (SSC) guidelines recommended administration of at least 30 mL/kg of crystalloid fluid within the first 3 hours for patients with sepsis-induced hypoperfusion, followed by hemodynamic-guided adjustment.Because many participants in these large trials had already received similar volumes before randomization, this dosage became associated with favorable outcomes. The 2021 SSC guideline retained this recommendation, though downgraded from a "strong" to a "weak" recommendation in the absence of new high-quality evidence.This highlights persistent uncertainty and the need for further research on optimal fluid type and strategy in sepsis resuscitation.

Increasing attention has been paid to microcirculation in recent years. While macrocirculatory parameters such as blood pressure may normalize after resuscitation, this does not necessarily indicate restoration of tissue-level perfusion.Persistent microcirculatory dysfunction may contribute to inadequate oxygen delivery and delayed organ recovery. Understanding how different fluid therapies influence both macro- and microcirculation is therefore crucial for optimizing outcomes.

Currently used resuscitation fluids include crystalloids and colloids. Crystalloids rapidly redistribute into the interstitial space and may exacerbate tissue edema-particularly in sepsis where capillary permeability is increased-potentially impairing microcirculatory flow.Colloids contain larger molecules that remain intravascular for longer periods, generating oncotic pressure and maintaining circulating volume more effectively, which may theoretically support microcirculatory perfusion and oxygen delivery. Clinically used colloids include albumin, hydroxyethyl starch (HES), and gelatin. Albumin is effective but costly and limited in availability. HES has fallen out of favor due to its association with kidney injury and increased mortality in sepsis.Gelatin, derived from bovine collagen hydrolysates, is now the only artificial colloid still recommended by guidelines for hypovolemia in sepsis patients.Nevertheless, high-quality randomized controlled evidence comparing gelatin with crystalloids in sepsis remains insufficient.

Based on this background, the present study focuses on balanced gelatin solution-a compound solution containing 4% succinylated gelatin in a balanced crystalloid carrier. We hypothesize that, compared with balanced crystalloid alone, balanced gelatin may better support hemodynamic stability through its colloid osmotic effect, more effectively correct fluid imbalance, improve microcirculatory perfusion, promote organ function recovery, and ultimately improve clinical outcomes. This randomized controlled trial is designed to rigorously test this hypothesis.

Patient and Public Involvement (PPIE)

During the protocol development stage, this study incorporated Patient and Public Involvement (PPIE). Three public contributors without medical backgrounds were invited to review the full protocol and informed consent form prior to study initiation. They provided feedback from the perspective of typical patients and family members. The main areas of concern included:

* The need for more accessible and patient-friendly language when describing the study background and objectives.
* Difficulty understanding the double-blind design, with recommendations to use analogies or simplified explanations.
* High concern regarding safety issues, including allergic reactions, kidney injury, and fluid-related adverse events, and a desire for clear descriptions of emergency procedures and contact information.
* Interest in treatment stability, postoperative supportive care needs, long-term complications, and follow-up arrangements.
* Questions regarding treatment-related costs, the exploratory nature of the intervention, and whether future protocol optimization is planned.
* Expectation that overall study results will be shared with participants after study completion.

Based on this feedback, the research team has revised and optimized the protocol background, the explanation of "double-blind" in the informed consent form, the safety management procedures, the follow-up plan, and the approach for disseminating study results. These adjustments aim to enhance the clarity, acceptability, and overall engagement of patient participants.

Study Objectives Primary Objective To evaluate the effectiveness of balanced gelatin solution in perioperative fluid management for septic patients undergoing emergency non-cardiac surgery, with emphasis on:reducing perioperative positive fluid balance；promoting hemodynamic stability；improving microcirculatory perfusion；and supporting organ function recovery and clinical outcomes.

Secondary Objective To assess the safety of balanced gelatin solution in this population, focusing on its effects on kidney function, coagulation status, and common postoperative complications.

Study Design This is a prospective, multicenter, randomized, double-blind, controlled clinical trial with an adaptive design incorporating sample size re-estimation. An initial sample size of 318 patients (159 per group) will be recruited, with an interim analysis after enrollment of 50% of participants to reassess the required sample size. Patients are randomized in a 1:1 ratio to receive either balanced gelatin or crystalloid solution (Ringer's acetate). Randomization is stratified by baseline blood lactate level (≤ 4 mmol/L vs > 4 mmol/L) using a central dynamic allocation system to ensure balance between groups.

Population Eligible patients are adults (≥18 years) with sepsis (per Sepsis-3 criteria) due to abdominal infection requiring emergency surgery. Inclusion requires a SOFA score ≥2 and lactate >2 mmol/L. Key exclusions include prior colloid use within 24 hours, expected death within 48 hours, advanced heart failure, severe ARDS, pre-existing renal replacement therapy, severe coagulopathy, liver failure, or allergy to gelatin.

Interventions All participants receive standardized anesthesia care. Intraoperative fluid therapy follows a goal-directed protocol guided by stroke volume monitoring. After randomization, patients in the intervention group receive balanced gelatin solution as the resuscitation fluid (maximum dose 30 mL/kg within 24 hours), while controls receive Ringer's acetate only. Both groups receive a baseline infusion of Ringer's acetate at 3 mL/kg/h during anesthesia. Vasoactive drugs are used according to predefined hemodynamic triggers. Postoperatively, the assigned fluid regimen is continued for 24 hours, after which fluid management follows routine clinical practice.

Endpoints

Primary endpoints include:

Cumulative fluid balance within 24 hours after surgery. Proportion of patients achieving hemodynamic stability within 24 hours. Secondary endpoints include kidney function, SOFA score dynamics, lactate clearance, need for vasopressors or renal replacement therapy, postoperative complications, ICU and hospital length of stay, and all-cause mortality at 28 and 90 days. Safety endpoints include pulmonary edema, arrhythmias, and acute kidney injury.

Follow-up Patients will be followed during hospitalization and by structured telephone interviews at day 28 and day 90. Follow-up assessments include survival, complications, and health-related quality of life using the EQ-5D-5L questionnaire.

Blinding and Oversight The study is double-blind: patients, treating clinicians, outcome assessors, and statisticians remain unaware of group allocation. Randomization and drug packaging are handled by independent, unblinded coordinators. Emergency unblinding is permitted only for patient safety. An independent Data and Safety Monitoring Board (DSMB) will oversee trial conduct and review adverse events.

Significance By directly comparing balanced gelatin with crystalloids in septic patients undergoing emergency abdominal surgery, this trial will provide critical evidence regarding the efficacy and safety of gelatin-based fluid resuscitation. Results are expected to inform perioperative fluid management strategies and contribute to guideline development in the management of sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Diagnosis of sepsis according to Sepsis-3 definition.
* Scheduled for emergency non-cardiac surgery under general anesthesia.
* Randomization and study intervention can be initiated before skin incision.
* Provision of written informed consent by patient or legal representative.

Exclusion Criteria:

* Cardiac surgery, neurosurgery, or procedures requiring cardiopulmonary bypass.
* Severe preexisting cardiac dysfunction (ejection fraction <30%, NYHA class IV).
* End-stage renal disease requiring chronic renal replacement therapy.
* Known severe hepatic failure (Child-Pugh C).
* Known allergy or contraindication to study fluids (gelatin solution or crystalloid solution).
* Pregnant or lactating women.
* Participation in another interventional trial within the past 30 days.
* Life expectancy <24 hours or decision to withhold/withdraw life-sustaining treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome 1: Net fluid balance within 24 hours after surgery | Intraoperative period and postoperative 24 hours
  Net fluid balance is defined as the difference between total infused volume and total output volume during surgery and the first 24 postoperative hours.
  Input volume includes all study fluids (balanced gelatin solution or acetate Ringer's), albumin, blood products, and maintenance crystalloid infusion. Excluded are solvent volumes <50 mL and non-therapeutic fluids such as irrigation or enteral/oral intake. Albumin is recorded in mL of solution administered. Blood product volumes are standardized: packed red blood cells 1 unit = 200 mL; plasma = actual volume; apheresis platelets 1 therapeutic dose = 250 mL; cryoprecipitate 1 unit = 25 mL (with center-specific adjustment allowed).
  Output volume includes intraoperative blood loss, urine output, and measurable drainage (thoracic, abdominal, nasogastric, etc.), excluding insensible or unmeasurable losses.
Primary Outcome 2: Proportion of patients achieving hemodynamic stability within 24 hours after surgery | Postoperative 24 hours
  Hemodynamic stability (HDS) is defined as meeting all of the following three criteria at postoperative 24 hours:
  1. Mean arterial pressure (MAP) ≥65 mmHg without vasopressor support, sustained ≥1 hour after discontinuation of vasopressors, with all subsequent MAP measurements ≥65 mmHg.
  2. Blood lactate ≤2 mmol/L, based on the most recent venous or arterial sample.
  3. Urine output ≥1 mL/kg/h, based on the average over the preceding 6 hours. The outcome measure is the percentage of patients in each group who fulfill all three criteria.

SECONDARY OUTCOMES:
Secondary Outcome 1.1: Intensity of study drug use within 24 hours after surgery | Randomization to postoperative 24 hours
  Cumulative volume of study drug administered from randomization to 24 hours postoperatively, standardized by ideal body weight (mL/kg).
Secondary Outcome 1.2: Blood product utilization rate within 24 hours after surgery | Randomization to postoperative 24 hours
  Proportion of patients receiving any blood product during the intervention period, regardless of type. Each patient is counted once even if multiple blood products are used.
Secondary Outcome 1.3: Vasopressor load within 24 hours after surgery | Randomization to postoperative 24 hours
  Vasopressor dose converted to norepinephrine-equivalent according to predefined equivalence table (norepinephrine:epinephrine:dopamine:phenylephrine:vasopressin = 1:1:0.01:0.01:0.02), normalized by ideal body weight and infusion time (μg/kg/min).
Secondary Outcome 1.4: Proportion of patients receiving inotropic drugs within 24 hours after surgery | Randomization to postoperative 24 hours
  Proportion of patients treated with any inotrope (dobutamine, milrinone, levosimendan, etc.) within 24 hours postoperatively.
Secondary Outcome 2.1: Intraoperative lactate reduction magnitude | Baseline to end of surgery
  Difference between baseline lactate and lactate at end of surgery (mmol/L).
Secondary Outcome 2.2: 24-hour lactate reduction magnitude | Baseline to postoperative 24 hours
  Difference between baseline lactate and lactate at 24 hours after surgery (mmol/L).
Secondary Outcome 2.3: Normalization rate of capillary refill time (CRT) at end of surgery | From baseline to end of surgery
  Proportion of patients with CRT ≤3 seconds at end of surgery, measured every 30 minutes from preoperative period to end of surgery using standardized glass-slide method.
Secondary Outcome 3.1: Proportion of patients with decrease in SOFA score at postoperative day 3 compared with baseline | Baseline (preoperative) to postoperative day 3
  SOFA (Sequential Organ Failure Assessment) score is used to evaluate dysfunction across six organ systems (respiratory, coagulation, hepatic, cardiovascular, renal, and central nervous system), with each system scored from 0 to 4 and a total score ranging from 0 to 24.
  In this study, SOFA scoring follows the updated SOFA-2 criteria, including standardized rules for handling sedation, intubation, and mortality.
  Improvement is defined as a decrease in the total SOFA score at postoperative day 3 compared with baseline (score difference > 0). If the SOFA score does not decrease or increases (difference ≤ 0), the patient is categorized as not improved.
Secondary Outcome 3.2: Proportion of patients with severe organ dysfunction within 3 days after surgery | Postoperative day 1 to day 3
  Severe organ dysfunction is defined as SOFA score ≥3 in any organ system (respiratory, coagulation, liver, cardiovascular, renal, CNS) at least once during POD1-3. Deaths are counted as maximum scores.
Secondary Outcome 3.3: Incidence of acute kidney injury within 3 days after surgery | Baseline to postoperative day 3
  Acute kidney injury (AKI) is defined according to KDIGO 2012 criteria, assessed at POD1, POD2, and POD3.
Secondary Outcome 3.4: Cumulative duration of renal replacement therapy within 28 days after surgery | Postoperative day 1 to day 28
  Total number of days on renal replacement therapy (CRRT, intermittent hemodialysis, or peritoneal dialysis) during the 28 days after surgery.
Secondary Outcome 3.5: Incidence of coagulopathy within 3 days after surgery | Baseline to postoperative day 3
  Coagulopathy is defined as PT prolongation >3 seconds from baseline or INR >1.5 at any time during POD1-3.
Secondary Outcome 3.6: Duration of ventilator-free time within 24 hours after surgery | Postoperative 24 hours
  Total hours without invasive or non-invasive mechanical ventilation in the first 24 hours postoperatively. Interruptions <1 hour are excluded.
Secondary Outcome 3.7: Duration of ventilator-free time within 7 days after surgery | Postoperative day 1 to day 7
  Total days without invasive or non-invasive mechanical ventilation during the first 7 postoperative days. Interruptions <1 day are excluded.
Secondary Outcome 3.8: Duration of vasopressor-free time within 24 hours after surgery | Postoperative 24 hours
  Total hours during which MAP ≥65 mmHg is maintained without vasopressor support, sustained ≥1 hour, within the first 24 hours.
Secondary Outcome 3.9: Duration of vasopressor-free time within 72 hours after surgery | Postoperative day 1 to day 3
  Total hours during which MAP ≥65 mmHg is maintained without vasopressor support, sustained ≥1 hour, within the first 72 hours.
Secondary Outcome 4.1: Length of ICU stay | From ICU admission to ICU discharge
  Number of calendar days spent in the intensive care unit after surgery.
Secondary Outcome 4.2: Length of total hospital stay | From hospital admission to discharge
  Number of calendar days from hospital admission to hospital discharge.
Secondary Outcome 5.1: All-cause mortality within 28 days after surgery | Postoperative day 1 to day 28
  Death from any cause within 28 days postoperatively.
Secondary Outcome 5.2: All-cause mortality within 90 days after surgery | Postoperative day 1 to day 90
  Death from any cause within 90 days postoperatively.

OTHER OUTCOMES:
Safety Outcome 1.1: Incidence of postoperative respiratory complications (ARDS) | Postoperative day 1 to day 7
  ARDS defined as PaO₂/FiO₂ ratio <200 at any arterial blood gas measurement within 7 days postoperatively. Patients without postoperative blood gas data are excluded. Deaths without ARDS evidence are counted as negative.
Safety Outcome 1.2: Incidence of postoperative cardiovascular complications (arrhythmias) | Postoperative day 1 to day 28
  New-onset arrhythmias within 28 days postoperatively, including supraventricular tachycardia, ventricular tachycardia, or atrial fibrillation/flutter. Multiple events in same patient count once.
Safety Outcome 1.3: Incidence of postoperative renal complications | Postoperative day 1 to day 28
  Defined as new renal dysfunction (serum creatinine ≥2× baseline) or need for renal replacement therapy (RRT) within 28 days after surgery. One patient counts once regardless of multiple events.
Safety Outcome 2.1: Health-related quality of life at postoperative day 90 | Postoperative day 90
  Health-related quality of life will be assessed at postoperative day 90 using the EuroQol 5-Dimension 5-Level questionnaire (EQ-5D-5L). The descriptive system covers five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression), each rated on 5 levels (1 = no problems, 5 = extreme problems). Responses are converted to a health state code (e.g., 21321), which is then mapped to a utility index score using the Chinese EQ-5D-5L value set (range: -0.391 to 1.000, where 1.000 = full health and values <0 represent states worse than death).
  In addition, participants will provide a self-rated health score on the EQ-VAS, a vertical visual analog scale ranging from 0 (worst imaginable health) to 100 (best imaginable health).
Exploratory Outcome 1.1: Minimum and maximum plasma osmolality during surgery | Intraoperative period (Tpre to T0)
  Plasma osmolality measured hourly from start of surgery (Tpre) to end of surgery (T0). Minimum and maximum values recorded.
Exploratory Outcome 1.2: Minimum pH value during surgery | Intraoperative period (Tpre to T0)
  Arterial blood gas pH measured hourly from Tpre to T0. Lowest recorded value used.
Exploratory Outcome 1.3: Central venous oxygen saturation (ScvO₂) before and after surgery | Preoperative (Tpre) and end of surgery (T0)
  ScvO₂ measured at Tpre and T0.
Exploratory Outcome 1.4: Central venous-to-arterial CO₂ gap (P(cv-a)CO₂) before and after surgery | Preoperative (Tpre) and end of surgery (T0)
  P(cv-a)CO₂ measured at Tpre and T0.
Exploratory Outcome 2.1: Sublingual microvascular flow index (MFI) | Preoperative (Tpre) and end of surgery (T0)
  Semi-quantitative assessment of microvascular flow using SDF or IDF imaging system, measured at Tpre and T0.
Exploratory Outcome 2.2: Perfused boundary region (PBR) | Preoperative (Tpre) and end of surgery (T0)
  Glycocalyx integrity marker, assessed by SDF or IDF imaging system, measured at Tpre and T0. Higher values indicate more severe damage.
Exploratory Outcome 2.3: Red blood cell flow velocity | Preoperative (Tpre) and end of surgery (T0)
  Quantitative assessment of RBC centerline velocity (μm/s) using particle tracking algorithm, measured at Tpre and T0.
Exploratory Outcome 3.1: Circulating biomarkers of early renal injury (NGAL, Cystatin C) | Preoperative (before anesthesia induction), end of surgery, postoperative day 1, postoperative day 2, and postoperative day 3
  Plasma neutrophil gelatinase-associated lipocalin (NGAL) and cystatin C concentrations will be measured to evaluate early renal injury.
Exploratory Outcome 3.2: Circulating biomarkers of coagulopathy (TAT, PAI-1) | Preoperative (before anesthesia induction), end of surgery, postoperative day 1, postoperative day 2, and postoperative day 3
  Plasma thrombin-antithrombin complex (TAT) and plasminogen activator inhibitor-1 (PAI-1) concentrations will be measured to assess coagulation function.
Exploratory Outcome 3.3: Circulating cardiac biomarker (NT-proBNP) | Preoperative (before anesthesia induction), end of surgery, postoperative day 1, postoperative day 2, and postoperative day 3
  Plasma N-terminal pro-B-type natriuretic peptide (NT-proBNP) concentration will be measured to assess cardiac stress.
Exploratory Outcome 3.4: Circulating inflammatory and immune biomarkers | Preoperative (before anesthesia induction), end of surgery, postoperative day 1, postoperative day 2, and postoperative day 3
  Plasma concentrations of procalcitonin (PCT), C-reactive protein (CRP/hs-CRP), interleukin-6 (IL-6), interleukin-10 (IL-10), and monocyte HLA-DR expression will be measured to evaluate systemic inflammation and immune response.
Exploratory Outcome 3.5: Circulating endothelial biomarkers (Syndecan-1, Ang-2) | Preoperative (before anesthesia induction), end of surgery, postoperative day 1, postoperative day 2, and postoperative day 3
  Plasma syndecan-1 and angiopoietin-2 concentrations will be measured to assess endothelial integrity and glycocalyx damage.
Exploratory Outcome 4.1: Incidence of postoperative gastrointestinal intolerance (POGI) | Postoperative day 1, postoperative day 3, and postoperative day 7
  Postoperative gastrointestinal intolerance is defined as an i-Feed score of 3-5 at postoperative day 1, day 3, or day 7, without ever reaching ≥6. Each patient will be counted once.
Exploratory Outcome 4.2: Incidence of postoperative gastrointestinal dysfunction (POGD) | Postoperative day 1, postoperative day 3, and postoperative day 7
  Postoperative gastrointestinal dysfunction is defined as an i-Feed score ≥6 at postoperative day 1, day 3, or day 7. Each patient will be counted once.

CONTACTS AND LOCATIONS:
Overall Officials: Changhong Miao, MD, Principal Investigator — Fudan University
Locations (9):
- China (9):
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjing, Tianjing
  - The Second Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital and Yuying Children's Hospital of Wenzhou Medical University (WMU), Wenzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided
At this time, the study team has not finalized an IPD sharing plan. This is a multicenter trial in critically ill patients; data governance, site ownership, and de-identification procedures are still under review. If sharing is pursued, it would be limited to a de-identified dataset sufficient to reproduce key findings-not the complete raw source data (e.g., free-text notes or imaging). Any decision will be guided by participant privacy, consent language, local/national regulations, and approvals by the sponsor/IRB/DSMB. Aggregate results will be reported in publications and on ClinicalTrials.gov.

REFERENCES:
- [Background] Knaus WA, Draper EA, Wagner DP, Zimmerman JE. APACHE II: a severity of disease classification system. Crit Care Med. 1985 Oct;13(10):818-29. PMID 3928249
- [Background] Hedrick TL, McEvoy MD, Mythen MMG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Postoperative Gastrointestinal Dysfunction Within an Enhanced Recovery Pathway for Elective Colorectal Surgery. Anesth Analg. 2018 Jun;126(6):1896-1907. doi: 10.1213/ANE.0000000000002742. PMID 29293183
- [Background] Lee DH, Dane MJ, van den Berg BM, Boels MG, van Teeffelen JW, de Mutsert R, den Heijer M, Rosendaal FR, van der Vlag J, van Zonneveld AJ, Vink H, Rabelink TJ; NEO study group. Deeper penetration of erythrocytes into the endothelial glycocalyx is associated with impaired microvascular perfusion. PLoS One. 2014 May 9;9(5):e96477. doi: 10.1371/journal.pone.0096477. eCollection 2014. PMID 24816787
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clin Pract. 2012;120(4):c179-84. doi: 10.1159/000339789. Epub 2012 Aug 7. No abstract available. PMID 22890468
- [Background] Vincent JL, Moreno R, Takala J, Willatts S, De Mendonca A, Bruining H, Reinhart CK, Suter PM, Thijs LG. The SOFA (Sepsis-related Organ Failure Assessment) score to describe organ dysfunction/failure. On behalf of the Working Group on Sepsis-Related Problems of the European Society of Intensive Care Medicine. Intensive Care Med. 1996 Jul;22(7):707-10. doi: 10.1007/BF01709751. No abstract available. PMID 8844239
- [Background] Chappell D, Jacob M, Hofmann-Kiefer K, Conzen P, Rehm M. A rational approach to perioperative fluid management. Anesthesiology. 2008 Oct;109(4):723-40. doi: 10.1097/ALN.0b013e3181863117. PMID 18813052
- [Background] Qureshi SH, Rizvi SI, Patel NN, Murphy GJ. Meta-analysis of colloids versus crystalloids in critically ill, trauma and surgical patients. Br J Surg. 2016 Jan;103(1):14-26. doi: 10.1002/bjs.9943. Epub 2015 Nov 2. PMID 26522616
- [Background] van der Heijden M, Verheij J, van Nieuw Amerongen GP, Groeneveld AB. Crystalloid or colloid fluid loading and pulmonary permeability, edema, and injury in septic and nonseptic critically ill patients with hypovolemia. Crit Care Med. 2009 Apr;37(4):1275-81. doi: 10.1097/CCM.0b013e31819cedfd. PMID 19242338
- [Background] Stockwell MA, Scott A, Day A, Riley B, Soni N. Colloid solutions in the critically ill. A randomised comparison of albumin and polygeline 2. Serum albumin concentration and incidences of pulmonary oedema and acute renal failure. Anaesthesia. 1992 Jan;47(1):7-9. doi: 10.1111/j.1365-2044.1992.tb01942.x. PMID 1536412
- [Background] Gondos T, Marjanek Z, Ulakcsai Z, Szabo Z, Bogar L, Karolyi M, Gartner B, Kiss K, Havas A, Futo J. Short-term effectiveness of different volume replacement therapies in postoperative hypovolaemic patients. Eur J Anaesthesiol. 2010 Sep;27(9):794-800. doi: 10.1097/EJA.0b013e32833b3504. PMID 20520555
- [Background] Tseng CH, Chen TT, Wu MY, Chan MC, Shih MC, Tu YK. Resuscitation fluid types in sepsis, surgical, and trauma patients: a systematic review and sequential network meta-analyses. Crit Care. 2020 Dec 14;24(1):693. doi: 10.1186/s13054-020-03419-y. PMID 33317590
- [Background] Marx G, Schindler AW, Mosch C, Albers J, Bauer M, Gnass I, Hobohm C, Janssens U, Kluge S, Kranke P, Maurer T, Merz W, Neugebauer E, Quintel M, Senninger N, Trampisch HJ, Waydhas C, Wildenauer R, Zacharowski K, Eikermann M. Intravascular volume therapy in adults: Guidelines from the Association of the Scientific Medical Societies in Germany. Eur J Anaesthesiol. 2016 Jul;33(7):488-521. doi: 10.1097/EJA.0000000000000447. No abstract available. PMID 27043493
- [Background] Brunkhorst FM, Engel C, Bloos F, Meier-Hellmann A, Ragaller M, Weiler N, Moerer O, Gruendling M, Oppert M, Grond S, Olthoff D, Jaschinski U, John S, Rossaint R, Welte T, Schaefer M, Kern P, Kuhnt E, Kiehntopf M, Hartog C, Natanson C, Loeffler M, Reinhart K; German Competence Network Sepsis (SepNet). Intensive insulin therapy and pentastarch resuscitation in severe sepsis. N Engl J Med. 2008 Jan 10;358(2):125-39. doi: 10.1056/NEJMoa070716. PMID 18184958
- [Background] Perner A, Haase N, Guttormsen AB, Tenhunen J, Klemenzson G, Aneman A, Madsen KR, Moller MH, Elkjaer JM, Poulsen LM, Bendtsen A, Winding R, Steensen M, Berezowicz P, Soe-Jensen P, Bestle M, Strand K, Wiis J, White JO, Thornberg KJ, Quist L, Nielsen J, Andersen LH, Holst LB, Thormar K, Kjaeldgaard AL, Fabritius ML, Mondrup F, Pott FC, Moller TP, Winkel P, Wetterslev J; 6S Trial Group; Scandinavian Critical Care Trials Group. Hydroxyethyl starch 130/0.42 versus Ringer's acetate in severe sepsis. N Engl J Med. 2012 Jul 12;367(2):124-34. doi: 10.1056/NEJMoa1204242. Epub 2012 Jun 27. PMID 22738085
- [Background] Guidet B, Martinet O, Boulain T, Philippart F, Poussel JF, Maizel J, Forceville X, Feissel M, Hasselmann M, Heininger A, Van Aken H. Assessment of hemodynamic efficacy and safety of 6% hydroxyethylstarch 130/0.4 vs. 0.9% NaCl fluid replacement in patients with severe sepsis: the CRYSTMAS study. Crit Care. 2012 May 24;16(3):R94. doi: 10.1186/cc11358. PMID 22624531
- [Background] De Backer D, Donadello K, Sakr Y, Ospina-Tascon G, Salgado D, Scolletta S, Vincent JL. Microcirculatory alterations in patients with severe sepsis: impact of time of assessment and relationship with outcome. Crit Care Med. 2013 Mar;41(3):791-9. doi: 10.1097/CCM.0b013e3182742e8b. PMID 23318492
- [Background] Bruno RR, Wollborn J, Fengler K, Flick M, Wunder C, Allgauer S, Thiele H, Schemmelmann M, Hornemann J, Moecke HME, Demirtas F, Palici L, Franz M, Saugel B, Kattan E, De Backer D, Bakker J, Hernandez G, Kelm M, Jung C. Direct assessment of microcirculation in shock: a randomized-controlled multicenter study. Intensive Care Med. 2023 Jun;49(6):645-655. doi: 10.1007/s00134-023-07098-5. Epub 2023 Jun 6. PMID 37278760
- [Background] Ince C. Hemodynamic coherence and the rationale for monitoring the microcirculation. Crit Care. 2015;19 Suppl 3(Suppl 3):S8. doi: 10.1186/cc14726. Epub 2015 Dec 18. PMID 26729241
- [Background] Evans L, Rhodes A, Alhazzani W, Antonelli M, Coopersmith CM, French C, Machado FR, Mcintyre L, Ostermann M, Prescott HC, Schorr C, Simpson S, Wiersinga WJ, Alshamsi F, Angus DC, Arabi Y, Azevedo L, Beale R, Beilman G, Belley-Cote E, Burry L, Cecconi M, Centofanti J, Coz Yataco A, De Waele J, Dellinger RP, Doi K, Du B, Estenssoro E, Ferrer R, Gomersall C, Hodgson C, Moller MH, Iwashyna T, Jacob S, Kleinpell R, Klompas M, Koh Y, Kumar A, Kwizera A, Lobo S, Masur H, McGloughlin S, Mehta S, Mehta Y, Mer M, Nunnally M, Oczkowski S, Osborn T, Papathanassoglou E, Perner A, Puskarich M, Roberts J, Schweickert W, Seckel M, Sevransky J, Sprung CL, Welte T, Zimmerman J, Levy M. Surviving sepsis campaign: international guidelines for management of sepsis and septic shock 2021. Intensive Care Med. 2021 Nov;47(11):1181-1247. doi: 10.1007/s00134-021-06506-y. Epub 2021 Oct 2. No abstract available. PMID 34599691
- [Background] Kuttab HI, Lykins JD, Hughes MD, Wroblewski K, Keast EP, Kukoyi O, Kopec JA, Hall S, Ward MA. Evaluation and Predictors of Fluid Resuscitation in Patients With Severe Sepsis and Septic Shock. Crit Care Med. 2019 Nov;47(11):1582-1590. doi: 10.1097/CCM.0000000000003960. PMID 31393324
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Dellinger RP. The Surviving Sepsis Campaign: Where have we been and where are we going? Cleve Clin J Med. 2015 Apr;82(4):237-44. doi: 10.3949/ccjm.82gr.15001. PMID 25955458
- [Background] Schorr CA, Zanotti S, Dellinger RP. Severe sepsis and septic shock: management and performance improvement. Virulence. 2014 Jan 1;5(1):190-9. doi: 10.4161/viru.27409. Epub 2013 Dec 11. PMID 24335487
- [Background] Levy MM, Rhodes A, Phillips GS, Townsend SR, Schorr CA, Beale R, Osborn T, Lemeshow S, Chiche JD, Artigas A, Dellinger RP. Surviving Sepsis Campaign: association between performance metrics and outcomes in a 7.5-year study. Crit Care Med. 2015 Jan;43(1):3-12. doi: 10.1097/CCM.0000000000000723. PMID 25275252
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Background] Mouncey PR, Osborn TM, Power GS, Harrison DA, Sadique MZ, Grieve RD, Jahan R, Harvey SE, Bell D, Bion JF, Coats TJ, Singer M, Young JD, Rowan KM; ProMISe Trial Investigators. Trial of early, goal-directed resuscitation for septic shock. N Engl J Med. 2015 Apr 2;372(14):1301-11. doi: 10.1056/NEJMoa1500896. Epub 2015 Mar 17. PMID 25776532
- [Background] ARISE Investigators; ANZICS Clinical Trials Group; Peake SL, Delaney A, Bailey M, Bellomo R, Cameron PA, Cooper DJ, Higgins AM, Holdgate A, Howe BD, Webb SA, Williams P. Goal-directed resuscitation for patients with early septic shock. N Engl J Med. 2014 Oct 16;371(16):1496-506. doi: 10.1056/NEJMoa1404380. Epub 2014 Oct 1. PMID 25272316
- [Background] ProCESS Investigators; Yealy DM, Kellum JA, Huang DT, Barnato AE, Weissfeld LA, Pike F, Terndrup T, Wang HE, Hou PC, LoVecchio F, Filbin MR, Shapiro NI, Angus DC. A randomized trial of protocol-based care for early septic shock. N Engl J Med. 2014 May 1;370(18):1683-93. doi: 10.1056/NEJMoa1401602. Epub 2014 Mar 18. PMID 24635773
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169